CLINICAL TRIAL: NCT01689415
Title: Pilot Study in Renal Denervation in Patients With Stroke and Uncontrolled Hypertension
Brief Title: Renal Denervation Hypertension After Stroke
Acronym: REHEARSE
Status: Terminated | Type: Observational
Why Stopped: Based on results from SYMPLICITY HTN-3
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Associate Research Professor, Consultant neurologist, Bispebjerg Hospital
Other Study IDs: H-4-2012-102
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Hypertension
Keywords: Renal nerve denervation
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is known, that hypertension is the major risk factor of stroke and recurrent stroke. Blood pressure reduction - together with antithrombotics - remain crucial in stroke prevention.

This pilot study will examine the effect of renal nerve denervation in patients with treatment resistant hypertension after ischemic stroke or DWI/DTI-verified stroke. With 24 hours blood pressure measurements the effect after renal nerve denervation is examined 1,3,6 and 12 months after the procedure.

DETAILED DESCRIPTION:
Radio frequent ablation is used to renal nerve denervation (RND) and is a new invasive method used in treatment for hypertensive patients, where the sympathetic nerves to the kidneys ablates. RND shows a significant reduction in the systolic and diastolic blood pressure in patients with treatment resistant hypertension.

The hypothesis is that RDN is able to reduce the blood pressure in patients with previous stroke and treatment resistant hypertension and thereby reduce the risk of a new stroke.

Aim of study:

1. To validate the reduction in blood pressure after RND in patients with stroke and treatment resistant hypertension compared to the results achieved in patients only with essential hypertension
2. To examine if this treatment is possible on patients after stroke (procedure related limitations and security of the patient)
3. To describe the effect of RND in the development of changes in the white matter over time

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Clinical verified stroke within the last year
* Treatment resistant hypertension at 150 mm Hg or higher systolic at consultation
* Modified Ranking between 0-2

Exclusion Criteria:

* Lack of informed consent
* Renal artery anatomy, which prevents the procedure
* Reno vascular disease
* Pacemaker
* Haemodynamic vascular occlusion or valve disease
* Pregnancy or women in the childbearing age
* Secondary hypertension
* Mean systolic blood pressure over 180 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the study population must be 18+ years old and have a clinical verified stroke within the last year and treatment resistant hypertension at 150 mm Hg or higher systolic at consultation. The patients Modified Ranking Scale must be between 0-2.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
24 hour blood pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, MD,Ph.D,DMSci, Principal Investigator — Bispebjerg Hospital - Department of neurology
Locations (1):
- Bispebjerg Hospital, Department of neurology, Copenhagen, Region H, Denmark

REFERENCES:
- [Background] Friday G, Alter M, Lai SM. Control of hypertension and risk of stroke recurrence. Stroke. 2002 Nov;33(11):2652-7. doi: 10.1161/01.str.0000033929.62136.6f. PMID 12411656
- [Background] van Gijn J. The PROGRESS Trial: preventing strokes by lowering blood pressure in patients with cerebral ischemia. Emerging therapies: critique of an important advance. Stroke. 2002 Jan;33(1):319-20. No abstract available. PMID 11779934
- [Background] Kaplan NM. Resistant hypertension. J Hypertens. 2005 Aug;23(8):1441-4. doi: 10.1097/01.hjh.0000174968.72212.ac. PMID 16003165
- [Background] Daugherty SL, Powers JD, Magid DJ, Tavel HM, Masoudi FA, Margolis KL, O'Connor PJ, Selby JV, Ho PM. Incidence and prognosis of resistant hypertension in hypertensive patients. Circulation. 2012 Apr 3;125(13):1635-42. doi: 10.1161/CIRCULATIONAHA.111.068064. Epub 2012 Feb 29. PMID 22379110
- [Background] Hornnes N, Larsen K, Boysen G. Blood pressure 1 year after stroke: the need to optimize secondary prevention. J Stroke Cerebrovasc Dis. 2011 Jan-Feb;20(1):16-23. doi: 10.1016/j.jstrokecerebrovasdis.2009.10.002. Epub 2010 Jun 17. PMID 21187254
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036